CLINICAL TRIAL: NCT04242589
Title: A Phase II Randomized Trial of Combined Radiotherapy and Vertebroplasty to Improve the Quality of Life of Patients With Painful Metastatic Localized Spinal Lesions
Brief Title: Trial of Combined Radiotherapy and Vertebroplasty for Patients With Painful Metastatic Spinal Lesions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0008
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Spinal Metastases
Keywords: Vertebroplasty; Vertebral Compression Fracture; Radiotherapy
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy (Active Comparator): Radiotherapy dose: 20 Gy/5 fractions/1 week or 8 Gy/1 fraction (at the discretion of the Radiation Oncologist)
  Interventions: Radiation: Radiotherapy
- Vertebroplasty + Radiotherapy (Experimental): Vertebroplasty followed by radiotherapy within 2-3 weeks
  Radiotherapy dose: 20 Gy/5 fractions/1 week or 8 Gy/1 fraction (at the discretion of the Radiation Oncologist)
  Interventions: Radiation: Radiotherapy; Procedure: Vertebropladty

INTERVENTIONS:
Radiation: Radiotherapy — External beam radiation therapy is a type of radiation therapy used for cancer treatment. A machine is used to aim high-energy rays from outside the body into tumor
  Other Names: External Beam Radiation Therapy
Procedure: Vertebropladty — Vertebroplasty is a procedure for stabilizing compression fractures in the spine. Bone cement is injected into vertebrae that have cracked or broken. The cement hardens, stabilizing the fractures and supporting your spine.
  Arms: Vertebroplasty + Radiotherapy

SUMMARY:
Since patients with spinal metastases are living longer, durable palliation with long-term tumor control are becoming increasingly important.

EBRT results in durable local control of bone metastasis. However, about 25 % of patients with spinal metastases only achieved complete pain relief following EBRT for a median duration of less than 4 months. This could be partly due to spinal instability. In addition, almost half of the patients who receive EBRT will subsequently develop VCFs . Hence, RT does not stabilize the spine secondary to VCFs and is not effective in preventing imminent VCFs. Vertebroplasty has rapidly reduced pain and improved function in patients with VCFs. However, vertebroplasty does not provide local tumor control similar to EBRT.

It is theorized that combining vertebroplasty with EBRT will stabilize the spine, relieve the pain, prevent imminent VCFs and minimize or avoid the need for opioids. It is hypothesized that combining a spine stabilization procedure such as vertebroplasty with RT will be the most effective management for patients with spinal metastases than RT alone for patients with spinal metastases. Combined vertebroplasty and radiotherapy is not a standard treatment option at present. This study is designed to quantify the advantage of adding vertebroplasty to radiotherapy for patients with spinal metastases. If the study is proven to be significant, it could become the standard of care for patients with spinal metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Participants capable of giving informed consent, or if appropriate, participants having an acceptable individual capable of giving consent on the participant's behalf
2. Patients must be 18 years of age or older
3. Spinal vertebral metastases confirmed by CT, MRI or bone scan.
4. Patients with painful (VAS of at least ≥ 2) vertebral spinal metastases in the thoracic and /or lumbar spine (not cervical).
5. Patients must be willing and able to comply with schedule visits, treatment plan, tests and other study procedures
6. Life expectancy > 6 months. Life expectancy will be evaluated by the study investigator both clinically and by using Linden model. Patient should be in the group B or C of the Linden model.
7. Patients with an ECOG score 0-2 or Karnofsky performance status of ≥ 60% will be eligible for enrolment (see appendix 1).
8. No prior EBRT to the target +/-1 vertebral body level
9. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause
10. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly (Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard) .
11. Females must not breastfeed during study treatment.
12. Male patients should agree to not donate sperm during study treatment.
13. Absence of any condition hampering compliance with study protocols and follow-up schedule; those conditions should be reviewed with the patient prior to trial registration

Exclusion Criteria

1. Patient cannot provide consent
2. Prior radiotherapy to the target +/-1 vertebral body level
3. Life expectancy < 6 months (assessed both clinically and using Linden model)
4. Karnofsky performance status of < 60%
5. Primary bone tumors
6. Plasmacytoma
7. Communicated fracture
8. Associated Impending cord compression or spinal cord compression
9. Epidural involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Pain Score based on the Visual Analog Scale | 1,3,6 and 12 months post treatment
  The primary end point is the improvement in pain score of at least 2 points (a decrease of 2 points) on the visual analogue Scale (VAS) without concurrent increase in opioids.
Improvement in Pain Score based on the Brief Pain Inventory | 1,3,6 and 12 months post treatment
  The primary end point is the improvement in pain score of at least 2 points (a decrease of 2 points) on the Brief Pain Inventory (BPI) without concurrent increase in opioids.

SECONDARY OUTCOMES:
Changes in back-specific physical functioning | 1,3,6 and 12 months post treatment
  The improvement in back-specific physical functioning is evaluated by the change in Roland-Morris disability questionnaire (RDQ) score.
Incidence of vertebral compression fractures post treatment. | Baseline, 6 months and 12 months
  The incidence of vertebral compression fractures will be evaluated by standing lateral spine radiographs of the thoracic and lumbar vertebrae.
Prospectively quantify pain response using the Visual Analog Scale | 1,3,6 and 12 months post treatment
  Pain response will be assessed by VAS and evaluated using a patient diary based on the International Bone Metastases Working Party Criteria. Based on intake of analgesics, the daily oral morphine equivalent dose (OMED) will be calculated.
Prospectively quantify pain response using the Brief Pain Inventory. | 1,3,6 and 12 months post treatment
  Pain response will be assessed by BPI and evaluated using a patient diary based on the International Bone Metastases Working Party Criteria. Based on intake of analgesics, the daily oral morphine equivalent dose (OMED) will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada